CLINICAL TRIAL: NCT04139434
Title: A Phase 1, Multicenter, Open-label, Dose-escalation Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Clinical Activity of Orally Administered LP-108 as Monotherapy and in Combination With Azacitidine in Subjects With Relapsed or Refractory Myelodysplastic Syndromes (MDS), Chronic Myelomonocytic Leukemia (CMML), or Acute Myeloid Leukemia (AML)
Brief Title: Dose-Escalation Study of Oral Administration of LP-108 as Monotherapy and in Combination With Azacitidine in Patients With Relapsed or Refractory MDS, CMML, or AML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Newave Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LP-108P
Record Dates: First submitted 2019-10-18; First posted 2019-10-25 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: AML/MDS; CMML; Relapse; Refractory Acute Lymphoblastic Leukemia; Relapse Leukemia; Relapsed Adult AML
Keywords: AML; MDS; CMML; relapse; refractory; LP-108
MeSH Terms: conditions — Recurrence; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Intervention Model Description: A classic "3+3" design will be used to establish dose-limiting toxicity (DLT), MTD, and RP2D.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Phase: LP-108 monotherapy (Experimental): Three to 6 subjects per treatment cohort will be assigned to receive sequentially higher oral doses of LP-108 on a once daily schedule for 28 days (a "Cycle") starting at a dose of 100 mg.
  Interventions: Drug: LP-108
- Dose Expansion Phase: LP-108 in combination with azacitidine (Experimental): Three to 6 subjects per treatment cohort will be assigned to receive sequentially higher oral doses of LP-108 on a once daily schedule for 28 days (a "Cycle") starting at a dose of 100 mg in combination with azacitidine at 75 mg/m2.
  Interventions: Drug: LP-108 and azacitidine

INTERVENTIONS:
Drug: LP-108 — For the dose escalation phase, LP-108 will be given once daily at the following dose levels: 100 mg QD, 200 mg QD, 400 mg QD, 600 mg QD, 800 mg QD, 1000 mg QD.
  Arms: Dose Escalation Phase: LP-108 monotherapy
Drug: LP-108 and azacitidine — For the dose escalation phase, LP-108 will be given once daily at the following dose levels: 100 mg QD, 200 mg QD, 400 mg QD, 600 mg QD, 800 mg QD, 1000 mg QD, with azacitidine at the standard dose of 75 mg/m2 on Day 1 - Day 7 of each 28-day cycle (weekly schedule) or on Days 1-5, 8, 9 of each 28-day cycle (5-2-2 schedule), according to institutional guidelines.
  Arms: Dose Expansion Phase: LP-108 in combination with azacitidine

SUMMARY:
A Phase 1, Multicenter, Open-label, Dose-escalation Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Clinical Activity of Orally Administered LP-108 as Monotherapy and in Combination with Azacitidine in Subjects with Relapsed or Refractory Myelodysplastic Syndromes (MDS), Chronic Myelomonocytic Leukemia (CMML), or Acute Myeloid Leukemia (AML)

DETAILED DESCRIPTION:
The primary objectives are to assess the safety and tolerability profile, determine the maximum tolerated dose (MTD), and/or the recommended Phase 2 dose (RP2D) of LP-108 administered daily as a single agent dosed orally and in combination with azacitidine at 75 mg/m2 in adult subjects with relapsed/refractory MDS/CMML/AML; to characterize the pharmacokinetics (PK) profile of LP-108 as monotherapy and in combination with azacitidine in adult subjects with relapsed/refractory MDS/CMML/AML.

Secondary objectives are to evaluate preliminary efficacy regarding the effect of LP-108 (monotherapy or combination therapy) on ORR for AML, MDS, CMML, PFS, DOR, and OS

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for study participation if the subject meets the following criteria:

* Eligible subject must have an advanced hematologic malignancy including:

  * MDS with refractory anemia with excess blasts (RAEB; subtype RAEB-1 or RAEB-2) as defined by World Health Organization (WHO) 2016 revised criteria and/or MDS with high- or very high-risk (risk score > 4.5) per the Revised International Prognostic Scoring System (IPSS-R) (Greenberg et al. 2012) that is relapsed or refractory to prior therapy for MDS, or the subject is intolerant to established therapy known to provide clinical benefit for their condition in the opinion of the Investigator; Or relapsed and/or refractory MDS subjects in whom the Investigators feel would benefit from Arm 2.
  * Relapsed and/or primary refractory AML as defined by WHO 2016 revised criteria; Or frontline older and/or unfit AML subjects in whom the Investigators feel would benefit from Arm 2.
  * CMML (with ≥ 5% blasts in bone marrow) as defined by WHO 2016 revised criteria that is relapsed and/or refractory and that, in the opinion of the Investigator, requires treatment or that has exhausted treatment options that would be considered standard of care.
  * Subject's prior therapies may include other BCL2 inhibitors and other HMA agents for Arm 2.
* Blast count ≤ 30 × 10^9 cells/L at the time of initiating investigational therapy (hydroxyurea is allowed to control blast count prior to and during therapy).
* Subject must have adequate coagulation, renal, and hepatic function.

  * Activated partial thromboplastin time and prothrombin time not to exceed 1.5 × the upper limit of normal (ULN);
  * Calculated creatinine clearance (Cr Cl) ≥ 30 mL/min using 24-hour CrCl OR Cockcroft-Gault formula (using actual body weight)
  * UK and EU only: Estimated glomerular filtration rate (GFR) ≥ 30 mL/min/1.73m2 using the modification of diet in renal disease (MDRD) equation.
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 ×ULN; bilirubin ≤ 1.5 × ULN (except subjects with Gilbert's Syndrome, who may have a bilirubin > 1.5 × ULN, per discussion between the Investigator and the Medical Monitor).
* Adequate cardiac function defined as: shortening fraction of ≥ 27% by echocardiogram, or ejection fraction of ≥ 50% by 2D echocardiogram without Doppler.

Exclusion Criteria:

A subject will not be eligible for study participation if he/she meets any of the following criteria.

* Subjects with a diagnosis of promyelocytic leukemia/retinoic acid receptor alpha (PML-RARA) or non-PML-RARA rearranged acute promyelocytic leukemia (APL).
* Subjects who have undergone hematopoietic stem cell transplantation (HSCT) within 60 days of the first dose of LP-108, or subjects on immunosuppressive therapy post-HSCT at the time of Screening, or with clinically significant graft-versus-host disease (GVHD). (Subjects in relapse after allogeneic transplantation must be off calcineurin inhibitors for at least 4 weeks. The use of topical steroids and/or up to 20 mg/day prednisone or equivalent systemic steroids for ongoing GVHD is permitted).
* Subject has received any of the following therapies within 14 days or 5 half-lives (whichever is shorter) prior to the first dose of study drug, or has not recovered to ≤ Grade 1 clinically significant adverse effect(s) of the previous therapy:

  * Any anti-cancer therapy including chemotherapy, hormonal therapy, biologic or immunotherapy, targeted small molecule agents, etc. (corticosteroid therapy < 20 mg/day prednisone equivalent for < 14 days at time of study treatment and hydroxyurea cytoreduction therapy according to institutional guidelines to treat disease associated symptoms are permitted).
  * Any investigational therapy.
  * There is 28-day washout period required for subject who have had prior CAR-T treatment if there is no evidence of cytokine release syndrome (CRS) or other adverse events related to the CAR-T treatment per discussion with the Medical Monitor.
* Subject has received the following medications or therapies within 7 days or 5 half-lives (whichever is shorter) prior to the first dose of study drug:

  * Cytochrome P450, family 3, subfamily A (CYP3A4) strong inhibitors (see Appendix 10 for strong CYP3A4 inhibitors). In Phase 1b of this trial, the criterion regarding CYP3A4 strong inhibitors will be removed at time of amendment of the trial when Phase 1b is to be initiated. The amendment will include recommendations on concomitant dosing of LP-108 and strong CYP3A4 inhibitors such as azole antifungal agents, PK monitoring for the initial weeks on study, as well as closer safety monitoring for subjects.
  * Strong CYP3A4 inducers such as rifampin, carbamazepine, phenytoin, and St. John's wort.
  * Inhibitors of P-glycoprotein (P-gp) and breast cancer resistance protein (BCRP) (see Appendix 11 for P gp and BCRP inhibitors).
  * Immunosuppressive drugs (equivalent to >10mg prednisone) for underlying autoimmune or rheumatologic conditions.
  * All statins as they could inhibit bilirubin uptake transporter OATP1B1 and OATP1B3 (the washout period should always be 5 half-lives) (see Appendix 11)
* Subject has baseline prolongation of the corrected QTc > 480 ms (calculated per Fridericia's formula [QTc = QT/RR (1/3)].
* Subject has a history of other malignancies other than the eligible hematologic malignancy within the past 1 year prior to study entry, with the exception of:

  * Subject with breast cancer or prostrate cancer on endocrine therapy with stable disease.
  * Adequately treated in situ carcinoma of the cervix uteri;
  * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin;
  * Previous malignancy confined and surgically resected (or treated with other
* Subject exhibits evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

  * Uncontrolled systemic infection (bacterial, fungal, viral)
  * Known active or poorly controlled human immunodeficiency virus or active hepatitis B or C infection
  * Unexplained fever > 38.5 °C during the Screening period or on their first day of study drug administration (at the discretion of the Investigator, if the fever is considered related to the subject's malignancy may be enrolled).
* Subjects with known and active central nervous system (CNS) involvement (radiographic or cytologic) at Screening; subjects with history of CNS involvement who have no symptoms suggestive of CNS disease and have had at least 2 successful lumbar punctures without cytologic evidence of leukemia may be included after discussion and approval of the Medical Monitor. (Evaluation of cerebrospinal fluid is only required if there is a clinical suspicion of CNS involvement by leukemia during screening in subjects without a history of CNS involvement).
* Subjects with immediate life-threatening, severe complications of leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation.
* Requires ongoing treatment with

  * Systemic acid-reducing agents including H-2-receptor antagonists and proton pump inhibitors
  * Sensitive CYP2C8 substrates (such as montelukast, pioglitazone, repaglinide, rosiglitazone) or CYP2C8 substrates with a narrow therapeutic index (e.g., amiodarone, fosphenytoin, paclitaxel, penprocoumon, phenytoin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | up to 13 cycles (one cycle has 4 weeks)
Recommended Phase 2 dose (RP2D) | up to 13 cycles (one cycle has 4 weeks)
The pharmacokinetic (PK) profile of LP-108: Maximum Plasma Concentration [Cmax] | At Cycle 1 Day 1 (24 h PK), Cycle 1 Day 8, Cycle 1 Day 15, Cycle 1 Day 22, Cycle 2 Day 1 (24 h PK)
The PK profile of LP-108: Area Under the Curve [AUC] | At Cycle 1 Day 1 (24 h PK), Cycle 1 Day 8, Cycle 1 Day 15, Cycle 1 Day 22, Cycle 2 Day 1 (24 h PK)
The PK profile of LP-108: Time at Maximum Concentration [Tmax] | At Cycle 1 Day 1 (24 h PK), Cycle 1 Day 8, Cycle 1 Day 15, Cycle 1 Day 22, Cycle 2 Day 1 (24 h PK)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) for AML | up to 13 cycles (one cycle has 4 weeks)
  Assessment will be based on revised recommendations of the ELN 2017.
ORR for MDS | up to 13 cycles (one cycle has 4 weeks)
  Assessment will be based on the proposed International Working Group 2006 criteria for MDS patients.
ORR for CMML | up to 13 cycles (one cycle has 4 weeks)
  Assessment will be based on international consortium proposal of uniform response criteria for myelodysplastic/myeloproliferative neoplasms (MDS/MPN) for CMML patients.
Progression-Free Survival (PFS) | up to 13 cycles (one cycle has 4 weeks)
  PFS is defined as the time from start of treatment until objective disease progression or death, whichever occurs first.
Duration of Response (DOR) | up to 13 cycles (one cycle has 4 weeks)
  DOR is for all subjects achieving an objective response.
Event-Free Survival (EFS) | up to 13 cycles (one cycle has 4 weeks)
  EFS is defined as the time from the start of LP-108 therapy until the earliest date of refractory disease or relapse.
Overall Survival (OS) | up to 13 cycles (one cycle has 4 weeks)
  Overall survival is defined as the time from treatment initiation until death from any cause.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - University of Michigan, Ann Arbor, Michigan
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State Comprehensive Cancer Center, Columbus, Ohio
  - MD Anderson Cancer Center, Huston, Texas
- Spain (3):
  - Institut Català d'oncologia - ICO Badalona, Badalona, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres, Cáceres
  - Instituto de Investigación Sanitaria La Fe, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No